CLINICAL TRIAL: NCT00775931
Title: Allogeneic Hematopoietic Stem Cell Transplantation For Severe Osteopetrosis
Brief Title: Allogeneic Transplantation For Severe Osteopetrosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MT2008-20; 0808M42261 (Other: Masonic Cancer Center, University of Minnesota)
Record Dates: First submitted 2008-10-16; First posted 2008-10-20 (Estimated); Results first posted 2019-07-31 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Severe Osteopetrosis
Keywords: osteopetrosis
MeSH Terms: conditions — Osteopetrosis | interventions — Cord Blood Stem Cell Transplantation; Alemtuzumab; Cyclophosphamide; Busulfan; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- marrow graft transplant conditioning (Active Comparator): Pre-transplant conditioning using Campath-1H, Busulfan, Fludarabine monophosphate, and total lymphoid irradiation followed by unrelated or matched related donor marrow graft transplantation (both peripheral blood and marrow) and a second CD34 cell infusion on Day 42.
  Interventions: Drug: Campath-1H; Radiation: Total Lymphoid Irradiation; Drug: Busulfan; Drug: Fludarabine monophosphate; Procedure: marrow graft transplantation
- cord blood transplant conditioning (Active Comparator): Pre-transplant conditioning using Campath-1H, Busulfan and Cyclophosphamide followed by unrelated umbilical cord blood transplantation and a second smaller portion cord blood graft infusion on Day 42.
  Interventions: Procedure: umbilical cord blood transplantation; Drug: Campath-1H; Drug: Cyclophosphamide; Drug: Busulfan

INTERVENTIONS:
Procedure: umbilical cord blood transplantation — Umbilical cord blood will be collected, processed and shipped according to existing protocols. 2 cord blood units will be utilized if available. The choice of units will be based on the HLA typing standards of the University of Minnesota Blood and Marrow Program. If 2 units are not available, a single unit may be used. If a single unit is used, the unit should provide at least 10 x 107 nucleated cells/kg recipient body weight.
  Other Names: UCBT
  Arms: cord blood transplant conditioning
Drug: Campath-1H — Campath-1H will be administered 0.3 mg/kg subcutaneously per day for three days starting on Day -21 through Day -19.
  Other Names: Alemtuzumab
Radiation: Total Lymphoid Irradiation — Dose 500 cGy via anteroposterior (AP) and posteroanterior(PA) fields (250 cGy AP and 250 cGy PA).
  Other Names: TLI
  Arms: marrow graft transplant conditioning
Drug: Cyclophosphamide — Cyclophosphamide (50 mg/kg/dose) will be given IV on day -4, -3, -2 and -1 over 2 hours. The total dose to be given over 4 days is 200 mg/kg for cord blood grafts-receiving patients only.
  Other Names: Cytoxan
  Arms: cord blood transplant conditioning
Drug: Busulfan — patients<12 kg: 1.1 mg/kg/dose IV every 6 hours for 8 doses total; patients >12 kg: 0.8 mg/kg/dose IV every 6 hours for 8 doses. on Day -8 to -7 for donor grafts-receiving patients, and on Day -9 to -6 for cord blood grafts-receiving patients.
  Other Names: Busulfex
Drug: Fludarabine monophosphate — Fludarabine (35 mg/m2 daily for 5 days, 175 mg/m2 total) will be administered IV over 30 minutes on days -6, -5, -4, -3, and -2 for donor grafts-receiving patients only.
  Other Names: Fludara
  Arms: marrow graft transplant conditioning
Procedure: marrow graft transplantation — Related donor marrow will be collected, processed and shipped according to existing protocols of the National Marrow Donor Program or other URD registry, with the goal of achieving a cell dose of ≥ 6.0 x 108 nucleated cells/kg. The proportion of cells that are CD34+ will be determined prior to the administration of the graft. This will allow a portion of the graft (2 x 106 CD34+ cells) to be frozen for a subsequent infusion on day +42.
  Other Names: HSCT
  Arms: marrow graft transplant conditioning

SUMMARY:
The purpose of this research is to explore what we believe may be a safer and more effective means of performing stem cell transplantation in patients with Osteopetrosis, using chemotherapy and radiation designed to bring about engraftment and lessen transplant mortality. Prior multi-institutional data in past studies found that approximately 30% of Osteopetrosis patients do not engraft. Therefore, in this study, we utilize a reduced intensity design of pre-transplant drugs to try to make transplants safer for this disease, as well as to provide a second infusion of stem cells in patients with matched related or unrelated donors.

DETAILED DESCRIPTION:
This revised transplant protocol will test the following: 1) the ability to achieve engraftment with the reduced intensity protocol and a second infusion of stem cells on day 42, 2) the mortality associated with transplant by day 100, 3) patient outcomes, based on differential imaging and biologic evaluations prior to transplantation and at designated points after transplantation (day 100, 6 months, 1, 2 and 5 years). Additional biologic studies will include microarray analysis, and evaluation of blood parameters and genes that may be important in the disease process. In older patients, studies to evaluation osteoclast differentiation and function will also be offered.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for transplantation under this protocol will be < or = 45 years of age, and will be diagnosed with severe osteopetrosis. This will be defined as having the following manifestations of the disease.

  1. Bones that are uniformly markedly dense based on skeletal survey
  2. No history that would suggest autosomal dominant inheritance
  3. Evidence of hematologic changes that are attributed to the underlying disease, including
* the need for ongoing transfusions, OR
* the presence of progressive anemia or thrombocytopenia, OR
* a white blood cell differential with a predominance of immature forms and evidence of extramedullary hematopoiesis, OR
* persistence of serious infectious complications that are thought to be due to the abnormal architecture of the bone that are resistant to surgical and medical interventions.

Exclusion Criteria:

* Patients >45 years of age
* Evidence of hepatic failure
* Pulmonary dysfunction sufficient to significantly increase the risk of transplant.
* Renal dysfunction with glomerular filtration rate (GFR) <30% of predicted.
* Cardiac compromise sufficient to substantially increase the risk of transplantation
* Severe, stable neurologic impairment.
* Human immunodeficiency virus (HIV) positivity.
* Pregnant or lactating females

Ages: 1 Day to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2008-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Orchard, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of MInnesota, Fairview, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cord Blood Transplant Conditioning: Pre-transplant conditioning using Campath-1H, Busulfan and Cyclophosphamide followed by unrelated umbilical cord blood transplantation and a second smaller portion cord blood graft infusion on Day 42.
  Campath-1H: Campath-1H will be administered 0.3 mg/kg subcutaneously per day for three days starting on Day -21 through Day -19.
  Busulfan: patients<12 kg: 1.1 mg/kg/dose IV every 6 hours for 8 doses total; patients >12 kg: 0.8 mg/kg/dose IV every 6 hours for 8 doses. on Day -8 to -7 for donor grafts-receiving patients, and on Day -9 to -6 for cord blood grafts-receiving patients.
  Cyclophosphamide: Cyclophosphamide (50 mg/kg/dose) will be given IV on day -4, -3, -2 and -1 over 2 hours. The total dose to be given over 4 days is 200 mg/kg for cord blood grafts-receiving
Period: Overall Study
Arm/Group | Marrow Graft Transplant Conditioning | Cord Blood Transplant Conditioning
Started | 6 | 1
Completed | 6 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Marrow Graft Transplant Conditioning | Cord Blood Transplant Conditioning | Total
Number analyzed (Participants) | 6 | 1 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 0 | 4
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Achieved Donor Cell Engraftment
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Marrow Graft Transplant Conditioning | Cord Blood Transplant Conditioning
Number analyzed (Participants) | 6 | 1
Participants | 5 | 0

2. Secondary Outcome: Transplant Related Mortality at 100 Days
Time Frame: day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Marrow Graft Transplant Conditioning | Cord Blood Transplant Conditioning
Number analyzed (Participants) | 6 | 1
Participants | 0 | 0

3. Secondary Outcome: Transplant Related Toxicity
Time Frame: Day 100 post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Marrow Graft Transplant Conditioning | Cord Blood Transplant Conditioning
Number analyzed (Participants) | 6 | 1
Participants | 3 | 1

4. Secondary Outcome: Incidence of Grade II - IV Acute Graft-versus-host Disease
Time Frame: by Day 100 after transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Marrow Graft Transplant Conditioning | Cord Blood Transplant Conditioning
Number analyzed (Participants) | 6 | 1
Participants | 2 | 0

ADVERSE EVENTS:
Arm/Group | Marrow Graft Transplant Conditioning | Cord Blood Transplant Conditioning
Serious Adverse Events (participants affected / at risk) | 3/6 | 0/1
Other Adverse Events (participants affected / at risk) | 6/6 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Marrow Graft Transplant Conditioning (N=6) | Cord Blood Transplant Conditioning (N=1)
Multi-Organ Failure (General disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 0
Acute Graft versus Host Disease (General disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Marrow Graft Transplant Conditioning (N=6) | Cord Blood Transplant Conditioning (N=1)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute Sinusitis (Infections and infestations) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Autoimmune Hemolytic Anemia (Blood and lymphatic system disorders) | 1 | 0
Bacterial Infection, Blood (Infections and infestations) | 4 | 0
Bacterial Infection, Respiratory (Infections and infestations) | 1 | 1
Bacterial Infection, Feces (Infections and infestations) | 1 | 1
Capillary Leak (Vascular disorders) | 1 | 0
Blood Clot in Bladder Wall (Blood and lymphatic system disorders) | 0 | 1
Requires Continuous Veno-Venous Hemofiltration, NOS (Renal and urinary disorders) | 1 | 0
Cystitis (Infections and infestations) | 2 | 0
Complete Heart Block (Cardiac disorders) | 1 | 0
Fungal Infection, Blood (Infections and infestations) | 2 | 0
Fungal Infection, Respiratory (Infections and infestations) | 3 | 1
Fungal Infection, Feces (Infections and infestations) | 0 | 1
Fungal Infection, Urine (Infections and infestations) | 1 | 0
Further Decompression of Lateral and Third Ventricles (Nervous system disorders) | 1 | 0
Requires Hemodialysis, NOS (Renal and urinary disorders) | 1 | 1
Hypertension (Vascular disorders) | 1 | 0
Hyperechogenic Renomegaly with Ascites (Renal and urinary disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Intracranial Hemorrhage (Nervous system disorders) | 1 | 0
Intraparenchymal Bleed (Nervous system disorders) | 1 | 0
Requires Intubation, NOS (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Large Splenic Infarct (Blood and lymphatic system disorders) | 0 | 1
Sinus Infection (Infections and infestations) | 1 | 0
Low Lung Volumes (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Obstruction of Left Proximal Internal Jugular Vein (Vascular disorders) | 1 | 0
Papilledema and Retinal Hemorrhages Leading to Blindness (Eye disorders) | 1 | 0
Partial Small Bowel Obstruction (Gastrointestinal disorders) | 1 | 0
Pericardial Effusion (Cardiac disorders) | 5 | 1
Placement of Epicardial Ventricular Pacing Wire (Cardiac disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Posterior Reversible Encephalopathy Syndrome (Nervous system disorders) | 1 | 0
Pulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Reactive Airway Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Seizure (Nervous system disorders) | 1 | 0
Small Bowel Ascites (Gastrointestinal disorders) | 0 | 1
Subconjunctival Hemorrhages (Eye disorders) | 1 | 0
Upper Respiratory Infection (Infections and infestations) | 1 | 0
Viral Infection, Blood (Infections and infestations) | 2 | 1
Viral Infection, Myocardium (Infections and infestations) | 1 | 0

LIMITATIONS AND CAVEATS:
Because the disease being treated on this study is rare, our intent was to only report these outcomes in context with other protocols. At some point in the future if we have enough patients we will analyze the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No